CLINICAL TRIAL: NCT04702750
Title: The Role of Context in Sleep-related Memory Reactivation in Humans: Reactivating Specific Memories During Sleep in Conjunction with a Suppression Context
Brief Title: Reactivating Specific Memories During Sleep in Conjunction with a Suppression Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Eitan Schechtman-Drayman, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00213443-C
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-11

CONDITIONS: Sleep; Consolidation
MeSH Terms: interventions — Odorants; Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Behavioral: Targeted memory reactivation (odors); Behavioral: Targeted memory reactivation (sounds)

INTERVENTIONS:
Behavioral: Targeted memory reactivation (odors) — I will unobtrusively and repeatedly present learning-related odors during sleep using an olfactometer. This method was shown to improve memory in various tasks. The odors will be presented in blocks with short breaks in-between. Odors will be pleasant as to not wake the participant up. The odors will be presented during non-rapid eye movement sleep (sleep stage 2 and slow wave sleep). The odors presented will be non-congruently associated with instructions in a previous learning task. This manipulation is within-subject - all participants will be exposed to all the odors during sleep, but odors will be associated with different instructions for each participant (counterbalanced).
Behavioral: Targeted memory reactivation (sounds) — I will unobtrusively and repeatedly present learning-related sounds during sleep using speakers. This method was shown to improve memory in various tasks. The sounds will be presented several seconds apart and the volume will be so adjusted as not to disturb the participant's sleep. The sounds will be presented during non-rapid eye movement sleep (sleep stage 2 and slow wave sleep). The sounds presented will be congruently related to the images in the previous learning task. This manipulation is within-subject - all participants will be exposed to sounds, but different specific sounds will be presented for each individual participant.

SUMMARY:
Forgetting is often perceived as the inability to retain information, but in fact at least some memory deterioration is due to active suppression processes, that are behaviorally adaptive. These active processes are thought to involve new, inhibitory learning, suggesting that sleep may serve to enhance them as it does other forms of learning. If this were the case, sleep may be harnessed to weaken non-adaptive memories in a manner that may be beneficial for healthy and clinical populations suffering from memory-related symptoms of disorders such as post-traumatic stress disorder (PTSD). To test this idea, this suggested nap study will incorporate specific memories in a suppression context during sleep monitored by encephalography (EEG). First, participants will take part in an item-based directed forgetting task, in which they will be exposed to different words, immediately followed by instructions to either remember the preceding word or not. The instructions will be conveyed using two distinct odors. In fact, the purpose of this first part would be to cement the associations of these odors with the instructions. Next, in an unrelated task, participants will learn the spatial locations of images on a screen. These images will be presented along with congruent sounds (e.g., cat - meow). During a subsequent nap, some of these sounds will be unobtrusively presented along with one of the two previously learned odors or along with a novel odor. In a final spatial-location test, memory for the images whose sounds were presented along with the "forget" odor during sleep is expected to be worse than for the images that were not cued. Memory for the locations of the images whose sounds were presented with one of the two other odors during sleep are expected to improve, possibly more so for the sounds presented with the "remember" odor relative to those presented with the novel odor. If successful, these results would be a first step towards interventions that may serve to selectively weaken memory during sleep.

DETAILED DESCRIPTION:
Each participant will be run in a single afternoon, which includes a 90-minute nap opportunity. Before the nap, participants will go through training and test sessions - and after it they will partake of final memory tests. Neural activity will be continuously monitored and recorded throughout the task using electrophysiological equipment. Breathing activity will also be measured.

This is a within-subjects study. The main manipulation is the unobtrusive presentation of sounds and odors during sleep, a technique called targeted memory reactivation (TMR). All participants will experience these stimuli, including all three odors, but the specific sounds each participant will hear will be different. Additionally, each of the three odors will be associated with specific instructions during wake (i.e., one odor instructing to remember a preceding word, another to forget it and one odor which will not be associated with any instructions). Odors will be counterbalanced across participants. The results will then be compared within participant, not between different groups or individuals. Appropriate statistical methods for such analyses include paired t-test and repeated measures analysis of variance. The choice of which sounds will be presented in conjunction with each of the odors (and which will not presented at all) for each participant will be made based on their performance in the pre-sleep test. This will be done in an attempt to balance pre-sleep scores between presented and unpresented stimuli to remove statistical noise. Both the participant and the experimenter will be blind to which sounds will be presented when, and the selection will be automatically made by the computer. This technique has been extensively used and has no known risks.

There are two main reasons that using a within-subject design reduces the required sample size. First, the lack of a between-subject independent variable intuitively requires less participants. Second, the level of statistical noise due to individual differences is reduced (i.e., because each participant is compared with their own scores). Previous TMR studies, which have found significant cuing effects, commonly used 20-25 participants. I plan to include at least 30 participants in this study, after omitting participants who could not complete the task and those who were not sufficiently cued during sleep. Having 30 participants will allow the use of more powerful statistical methods (in accordance with the common rule of thumb derived from the central limit theorem, which states that means based on sample sizes of more than 30 participants can be assumed to follow a normal distribution). My main interest in this study is the suppression TMR effect. It is hard to estimate the effect size of this detrimental effect, but it may be somewhat smaller than the typical TMR effect for spatial learning memories (Hedge's g = 0.39 based on a recent meta-analysis). To be on the safe side, I included a higher sample size. It is important to note that even if this benefit will be of a smaller magnitude, it will still be indicative of the potential for weakening memories during sleep. Aiming at a sample size of at least 30 participants and assuming an omission rate of 80%, I therefore plan to have 38 participants altogether.

Here is a brief summary of the procedure:

Stimuli: Three distinct odors which are equally arousing and pleasant will be used, for this study. A set of 100 nouns will be used to train participants on the directed forgetting task (see below). Finally, 60 images of objects or animals will be used, each with a unique 2D position on a circular grid presented on the screen.

Training: Participants will first participate in an item-based directed forgetting task. They will be shown a series of words and instructed, after every word, whether they should commit it to memory or not. The instructions will be delivered using two odors: one signaling to remember the last word (presented after 50 of the words) and the other to forget (presented after the other 50 words). To ensure that subjects use the odor in a time-locked manner, they will be instructed when they should sniff following each word's presentation (i.e., there will be an on-screen countdown culminating with the odor presentation and the instruction to sniff).

It should be noted that in my previous study, I had two suppression sounds, each associated with a different group, whereas here I only have one suppression odor. The justification for this is that in the previous study, sounds were associated with both the instructions and individual items. Here, I avoid this complexity, as each item has its own sound and the odors are used exclusively to convey suppression instructions. The interaction between odors and sounds in my study should achieve the desired suppression effect. Therefore, the design is more similar to the one used by Simon and colleagues, which used a single forget cue.

After this task, an unrelated spatial-learning task will begin. Participants will have to learn to position 60 images on a 2D circular grid. The task will be divided into 4 blocks, each beginning with exposure to the image locations, followed by positioning trials in which participants will have to place the items in their correct positions. Participants are expected to learn using feedback and will continue until reaching a learning criterion. Importantly, each image will be paired with a distinct, congruent sound during learning (e.g., cat - meow).

Pre-sleep test: After training, participants will be tested on their spatial-memory of all images with no feedback or sounds.

Sleep: Next, during NREM (non-rapid eye movement) sleep, I will unobtrusively present 75% of the image-related sounds from the latter task: 25% will be presented in the context of the "forget" odor; 25% will be presented in the context of the "remember" odor; and 25% will be presented in the context of a novel odor. The remaining 25% of sounds will not be presented during sleep. To avoid contamination between odors, I will use a block design (i.e., odors will be continuously presented, interspersed with sounds) with clean air breaks between blocks. Blocks will be ~20 seconds long to avoid odor habituation, and will be followed by a 20-second period during which clean air will be delivered. In each ~20 second block, 4 sounds will be presented. Using these setting, it should take approximately 7.5 minutes to cue all 45 sounds once.

Post-sleep test: At least 10 minutes after the end of the nap, participants will undergo a test identical to the pre-sleep one. Immediately after, they will be tested on the odor-instructions associations. Participants will then be thanked, debriefed, paid and dismissed.

ELIGIBILITY:
Inclusion Criteria:

---

Exclusion Criteria:

Participants with a history of neurological disorders or of sleep disorders will be excluded.

Participants who do not believe they would be able to fall asleep in the lab will be excluded.

Participants with severe asthma requiring hospitalization for treatment, history of significant food or non-food allergy, presence of known smell, taste or ear-nose-throat disorder, or a history of sinusitis or allergic rhinitis will be excluded.

Participants who are certain they breathe through their mouths during sleep and those who snore (and therefore likely breathe through their mouths as well) will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in error rates between pre- and post-sleep for the different conditions | Approximately 15 minutes before sleep onset and approximately 15 minutes after sleep offset within the same experimental session
  The correct location of an image is compared with the position in which the participant has placed it. Measured in pixels on a computer screen.
Modulation of EEG spectral power following sound/odor presentation | During sleep within the experimental session, assessed up to 1.5 hours
  Power modulations within the sigma (12-16 Hz), theta (4-8 Hz) and delta (0.5-4 Hz) ranges immediately following sound onset or at the first sniff after odor delivery. Measured across different EEG channels.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuroscience Lab - Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No